CLINICAL TRIAL: NCT02437903
Title: Open Label, Single-center Study, Evaluating the Efficacy and Safety of JUVÉDERM VOLUMA™ XC for the Facial Temporal Regions
Brief Title: Open Label Study Evaluating the Efficacy and Safety of JUVÉDERM VOLUMA™ XC for the Facial Temporal Regions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baumann Cosmetic and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Voluma Temporal 2014
Record Dates: First submitted 2015-04-30; First posted 2015-05-08 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-01

CONDITIONS: Aging
Keywords: voluma temporal, facial, volume loss
MeSH Terms: conditions — Facies

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (1):
- JUVÉDERM VOLUMA™ XC (Other): Subjects will be injected with JUVÉDERM VOLUMA™ XC to their right and left facial temporal regions at the baseline visit.
  Interventions: Device: JUVÉDERM VOLUMA™ XC

INTERVENTIONS:
Device: JUVÉDERM VOLUMA™ XC — Subjects will receive up to 4, 1mL syringes of JUVÉDERM VOLUMA™ XC for their initial injection and a maximum of 6, 1mL syringes of JUVÉDERM VOLUMA™ XC for the study. Subjects will undergo one touch-up injection approximately 2 weeks post initial treatment, and will continue to be evaluated at month 1, month 3, month 6, month 9, and month 12.
  Other Names: Injectable Dermal Filler

SUMMARY:
This study is to determine the efficacy and safety of JUVÉDERM VOLUMA™ XC when used in the facial temporal regions based on the change in the score of the investigator's Temporal. This study will be an open label, single center study.

DETAILED DESCRIPTION:
Volume deficit in the temporal area (the side of the forehead) of the face is a common sign of aging.

JUVÉDERM VOLUMA™ XC is a dermal filler, which was FDA-approved in October 2013 for the improvement and correction of age-related volume deficit in the mid-face area.

JUVÉDERM VOLUMA™ XC is a gel implant composed of 20 mg/mL hyaluronic acid (HA) formulation, produced by Streptococcus equi bacteria, and 0.3 w/w lidocaine. JUVÉDERM VOLUMA™ XC is a clear, sterile, and biodegradable gel indicated for subcutaneous and/or supraperiosteal injection.

JUVÉDERM VOLUMA™ XCwill be injected in the temple area and subjects will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to read and sign the informed consent and other study documents.
* Treating investigator's score of 3, 4, or 5 on the Temporal Fossa Rating Scale.
* Written informed consent has been obtained prior to any study-related procedures.
* Written Authorization for Use and Release of Health and Research Study Information has been signed.
* Ability to follow study instructions and complete study assessment tools including the subject diary
* Female patients of childbearing potential must have a negative urine pregnancy test result and not be lactating.
* Likely to complete all required visits with no plans to move from Miami in the next 12 months
* Agree to not undergo other treatments or cosmetic procedures in the treatment area during the study such as facial laser treatments, botulinum toxin, hyaluronic acid injections, subcutaneous fat injections, any other permanent or semi-permanent facial fillers.

Exclusion Criteria:

* Any uncontrolled systemic disease
* History of any of the following conditions: vision loss not corrected by lenses or LASIX surgery; glaucoma, retinal detachment, macular degeneration, history of multiple sclerosis or optic neuritis, or any uncontrolled eye disease.
* Have a history of severe allergic/anaphylactic reactions or multiple allergies.
* Conditions within the treatment area including acne, scarring, acute lupus erythematosus, dermatitis, or melasma.
* Females planning to become pregnant, are pregnant, or are breast-feeding.
* History or current evidence of drug or alcohol abuse within 12 months prior to the screening visit
* Have severe thin skin, in the treatment area as determined by the PI.
* Have undergone temporary facial dermal filler injections with hyaluronic acid-based fillers within 12 months in the treatment area. Have had neuromodulator injections, mesotherapy, or resurfacing (laser or other ablative or non-ablative procedures) within 5 months prior to entry in the study or be planning to undergo any of these procedures at any time during the study.
* Have undergone facial plastic surgery (with the exception of rhinoplasty or a brow lift), tissue grafting, or tissue augmentation with silicone, fat, or other permanent or semi-permanent dermal fillers or be planning to undergo any of these procedures affecting the treatment area, at any time during the study.
* Unwilling to undergo injections in the temple area.
* Have a history of migraines or frequent headaches, as determined by the PI.
* Have blindness or partial vision loss in either eye.
* Have received any other therapy, which, in the opinion of the investigator, could interfere with safety or efficacy evaluations.
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study.
* Patient who has a condition or is in a situation that, in the investigator's opinion, may put the patient at significant risk, or may significantly interfere with the patient's participation in the study.
* Have received anti-coagulation, anti-platelet, or thrombolytic medications (e.g.,warfarin), anti-inflammatory drugs (NSAIDs, e.g., aspirin, ibuprofen), or other substances known to increase coagulation time from 10 days pre- to 3 days post injection. A wash out period of 10 days is allowed.
* Have undergone immunosuppressive therapy, chemotherapy, biologics or systemic corticosteroids within 3 months prior to each study visit.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08-07 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie S Baumann, MD,CPI, Principal Investigator — Baumann Cosmetic and Research Institute
Locations (1):
- Baumann Cosmetic and Research Institute, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- JUVÉDERM VOLUMA™ XC: Subjects will be injected with JUVÉDERM VOLUMA™ XC to their right and left facial temporal regions at the baseline visit.
  JUVÉDERM VOLUMA™ XC: Subjects will receive up to 4, 1mL syringes of JUVÉDERM VOLUMA™ XC for their initial injection and a maximum of 6, 1mL syringes of JUVÉDERM VOLUMA™ XC for the study. Subjects will undergo one touch-up injection approximately 2 weeks post initial treatment, and will continue to be evaluated at month 1, month 3, and month 6.
Period: Overall Study
Arm/Group | JUVÉDERM VOLUMA™ XC
Started | 30
Completed | 25
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | JUVÉDERM VOLUMA™ XC
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Frontal Temporal Fossa Rating Scale
Description: Graded severity of the temporal line of the frontal bone (TLFB) using the Frontal Temporal Fossa Rating Scale: (these will have a picture assigned to each score.
Time Frame: Baseline, Month 1, Month 3, Month 6, Month 9, and Month 12
Population: All subjects with data for for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | JUVÉDERM VOLUMA™ XC
Number analyzed (Participants) | 30
Participants
  Temporal Fossa Rating Scale at Baseline: Severe Concavity | 10
  Temporal Fossa Rating Scale at Baseline: Moderate Concavity | 13
  Temporal Fossa Rating Scale at Baseline: Mild Concavity | 7
  Temporal Fossa Rating Scale at Baseline: Flat | 0
  Temporal Fossa Rating Scale at Baseline: Convexity | 0
  Temporal Fossa Rating Scale at Month 1: number analyzed (Participants) | 29
  Temporal Fossa Rating Scale at Month 1: Severe Concavity | 0
  Temporal Fossa Rating Scale at Month 1: Moderate Concavity | 0
  Temporal Fossa Rating Scale at Month 1: Mild Concavity | 1
  Temporal Fossa Rating Scale at Month 1: Flat | 27
  Temporal Fossa Rating Scale at Month 1: Convexity | 1
  Temporal Fossa Rating Scale at Month 3: number analyzed (Participants) | 26
  Temporal Fossa Rating Scale at Month 3: Severe Concavity | 0
  Temporal Fossa Rating Scale at Month 3: Moderate Concavity | 0
  Temporal Fossa Rating Scale at Month 3: Mild Concavity | 4
  Temporal Fossa Rating Scale at Month 3: Flat | 22
  Temporal Fossa Rating Scale at Month 3: Convexity | 0
  Temporal Fossa Rating Scale at Month 6: number analyzed (Participants) | 26
  Temporal Fossa Rating Scale at Month 6: Severe Concavity | 0
  Temporal Fossa Rating Scale at Month 6: Moderate Concavity | 0
  Temporal Fossa Rating Scale at Month 6: Mild Concavity | 8
  Temporal Fossa Rating Scale at Month 6: Flat | 18
  Temporal Fossa Rating Scale at Month 6: Convexity | 0
  Temporal Fossa Rating Scale at Month 9: number analyzed (Participants) | 25
  Temporal Fossa Rating Scale at Month 9: Severe Concavity | 0
  Temporal Fossa Rating Scale at Month 9: Moderate Concavity | 2
  Temporal Fossa Rating Scale at Month 9: Mild Concavity | 2
  Temporal Fossa Rating Scale at Month 9: Flat | 21
  Temporal Fossa Rating Scale at Month 9: Convexity | 0
  Temporal Fossa Rating Scale at Month 12: number analyzed (Participants) | 25
  Temporal Fossa Rating Scale at Month 12: Severe Concavity | 0
  Temporal Fossa Rating Scale at Month 12: Moderate Concavity | 0
  Temporal Fossa Rating Scale at Month 12: Mild Concavity | 5
  Temporal Fossa Rating Scale at Month 12: Flat | 20
  Temporal Fossa Rating Scale at Month 12: Convexity | 0

2. Secondary Outcome: Investigator's Satisfaction With the Appearance of the Temporal Regions
Description: Graded level of satisfaction with the current appearance of the temporal region making certain that the investigator is looking at the patient's right side and not the investigator's right side.
Time Frame: Baseline, Month 1, Month 3, Month 6, Month 9, and Month 12
Population: All subjects with data for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | JUVÉDERM VOLUMA™ XC
Number analyzed (Participants) | 30
Participants
  Investigator's Satisfaction at Baseline: Very Satisfied | 0
  Investigator's Satisfaction at Baseline: Moderately Satisfied | 0
  Investigator's Satisfaction at Baseline: Somewhat Satisfied | 0
  Investigator's Satisfaction at Baseline: Neither | 0
  Investigator's Satisfaction at Baseline: Somewhat Dissatisfied | 6
  Investigator's Satisfaction at Baseline: Moderately Dissatisfied | 12
  Investigator's Satisfaction at Baseline: Very Dissatisfied | 12
  Investigator's Satisfaction at Month 1: number analyzed (Participants) | 29
  Investigator's Satisfaction at Month 1: Very Satisfied | 24
  Investigator's Satisfaction at Month 1: Moderately Satisfied | 4
  Investigator's Satisfaction at Month 1: Somewhat Satisfied | 0
  Investigator's Satisfaction at Month 1: Neither | 0
  Investigator's Satisfaction at Month 1: Somewhat Dissatisfied | 0
  Investigator's Satisfaction at Month 1: Moderately Dissatisfied | 0
  Investigator's Satisfaction at Month 1: Very Dissatisfied | 1
  Investigator's Satisfaction at Month 3: number analyzed (Participants) | 26
  Investigator's Satisfaction at Month 3: Very Satisfied | 23
  Investigator's Satisfaction at Month 3: Moderately Satisfied | 3
  Investigator's Satisfaction at Month 3: Somewhat Satisfied | 0
  Investigator's Satisfaction at Month 3: Neither | 0
  Investigator's Satisfaction at Month 3: Somewhat Dissatisfied | 0
  Investigator's Satisfaction at Month 3: Moderately Dissatisfied | 0
  Investigator's Satisfaction at Month 3: Very Dissatisfied | 0
  Investigator's Satisfaction at Month 6: number analyzed (Participants) | 26
  Investigator's Satisfaction at Month 6: Very Satisfied | 18
  Investigator's Satisfaction at Month 6: Moderately Satisfied | 7
  Investigator's Satisfaction at Month 6: Somewhat Satisfied | 0
  Investigator's Satisfaction at Month 6: Neither | 0
  Investigator's Satisfaction at Month 6: Somewhat Dissatisfied | 1
  Investigator's Satisfaction at Month 6: Moderately Dissatisfied | 0
  Investigator's Satisfaction at Month 6: Very Dissatisfied | 0
  Investigator's Satisfaction at Month 9: number analyzed (Participants) | 25
  Investigator's Satisfaction at Month 9: Very Satisfied | 19
  Investigator's Satisfaction at Month 9: Moderately Satisfied | 3
  Investigator's Satisfaction at Month 9: Somewhat Satisfied | 1
  Investigator's Satisfaction at Month 9: Neither | 0
  Investigator's Satisfaction at Month 9: Somewhat Dissatisfied | 0
  Investigator's Satisfaction at Month 9: Moderately Dissatisfied | 2
  Investigator's Satisfaction at Month 9: Very Dissatisfied | 0
  Investigator's Satisfaction at Month 12: number analyzed (Participants) | 25
  Investigator's Satisfaction at Month 12: Very Satisfied | 16
  Investigator's Satisfaction at Month 12: Moderately Satisfied | 5
  Investigator's Satisfaction at Month 12: Somewhat Satisfied | 3
  Investigator's Satisfaction at Month 12: Neither | 0
  Investigator's Satisfaction at Month 12: Somewhat Dissatisfied | 1
  Investigator's Satisfaction at Month 12: Moderately Dissatisfied | 0
  Investigator's Satisfaction at Month 12: Very Dissatisfied | 0

3. Other Pre Specified Outcome: Subject's Satisfaction With Temple Appearance
Description: Subject's Satisfaction with Temple Appearance
Time Frame: Baseline, month 1, month 3, month 6, month 9, and Month 12
Population: All subjects with data for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | JUVÉDERM VOLUMA™ XC
Number analyzed (Participants) | 30
Participants
  Subject's Satisfaction at Baseline: Very Satisfied | 0
  Subject's Satisfaction at Baseline: Moderately Satisfied | 0
  Subject's Satisfaction at Baseline: Somewhat Satisfied | 0
  Subject's Satisfaction at Baseline: Neither | 2
  Subject's Satisfaction at Baseline: Somewhat Dissatisfied | 10
  Subject's Satisfaction at Baseline: Moderately Dissatisfied | 9
  Subject's Satisfaction at Baseline: Very Dissatisfied | 9
  Subject's Satisfaction at Month 1: number analyzed (Participants) | 29
  Subject's Satisfaction at Month 1: Very Satisfied | 18
  Subject's Satisfaction at Month 1: Moderately Satisfied | 9
  Subject's Satisfaction at Month 1: Somewhat Satisfied | 1
  Subject's Satisfaction at Month 1: Neither | 0
  Subject's Satisfaction at Month 1: Somewhat Dissatisfied | 0
  Subject's Satisfaction at Month 1: Moderately Dissatisfied | 0
  Subject's Satisfaction at Month 1: Very Dissatisfied | 1
  Subject's Satisfaction at Month 3: number analyzed (Participants) | 26
  Subject's Satisfaction at Month 3: Very Satisfied | 21
  Subject's Satisfaction at Month 3: Moderately Satisfied | 3
  Subject's Satisfaction at Month 3: Somewhat Satisfied | 2
  Subject's Satisfaction at Month 3: Neither | 0
  Subject's Satisfaction at Month 3: Somewhat Dissatisfied | 0
  Subject's Satisfaction at Month 3: Moderately Dissatisfied | 0
  Subject's Satisfaction at Month 3: Very Dissatisfied | 0
  Subject's Satisfaction at Month 6: number analyzed (Participants) | 26
  Subject's Satisfaction at Month 6: Very Satisfied | 15
  Subject's Satisfaction at Month 6: Moderately Satisfied | 7
  Subject's Satisfaction at Month 6: Somewhat Satisfied | 3
  Subject's Satisfaction at Month 6: Neither | 1
  Subject's Satisfaction at Month 6: Somewhat Dissatisfied | 0
  Subject's Satisfaction at Month 6: Moderately Dissatisfied | 0
  Subject's Satisfaction at Month 6: Very Dissatisfied | 0
  Subject's Satisfaction at Month 9: number analyzed (Participants) | 25
  Subject's Satisfaction at Month 9: Very Satisfied | 13
  Subject's Satisfaction at Month 9: Moderately Satisfied | 6
  Subject's Satisfaction at Month 9: Somewhat Satisfied | 4
  Subject's Satisfaction at Month 9: Neither | 1
  Subject's Satisfaction at Month 9: Somewhat Dissatisfied | 0
  Subject's Satisfaction at Month 9: Moderately Dissatisfied | 0
  Subject's Satisfaction at Month 9: Very Dissatisfied | 1
  Subject's Satisfaction at Month 12: number analyzed (Participants) | 25
  Subject's Satisfaction at Month 12: Very Satisfied | 14
  Subject's Satisfaction at Month 12: Moderately Satisfied | 5
  Subject's Satisfaction at Month 12: Somewhat Satisfied | 3
  Subject's Satisfaction at Month 12: Neither | 1
  Subject's Satisfaction at Month 12: Somewhat Dissatisfied | 1
  Subject's Satisfaction at Month 12: Moderately Dissatisfied | 0
  Subject's Satisfaction at Month 12: Very Dissatisfied | 1

4. Other Pre Specified Outcome: Subject Self-Perception of Age
Description: Subjects perception of age when the subject looks at his/her right and left temples
Time Frame: Baseline, month 1, month 3, month 6, month 9, and Month 12
Population: All subjects with data for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | JUVÉDERM VOLUMA™ XC
Number analyzed (Participants) | 30
Participants
  Subjects perception of age at Baseline: Same or Older | 23
  Subjects perception of age at Baseline: 1-5 Years Younger | 4
  Subjects perception of age at Baseline: 6-10 Years Younger | 3
  Subjects perception of age at Baseline: 11-15 Years Younger | 0
  Subjects perception of age at Baseline: 16+ Years Younger | 0
  Subjects perception of age at Baseline: Returned to Baseline | 0
  Subjects perception of age at Month 1: number analyzed (Participants) | 29
  Subjects perception of age at Month 1: Same or Older | 5
  Subjects perception of age at Month 1: 1-5 Years Younger | 14
  Subjects perception of age at Month 1: 6-10 Years Younger | 9
  Subjects perception of age at Month 1: 11-15 Years Younger | 1
  Subjects perception of age at Month 1: 16+ Years Younger | 0
  Subjects perception of age at Month 1: Returned to Baseline | 0
  Subjects perception of age at Month 3: number analyzed (Participants) | 26
  Subjects perception of age at Month 3: Same or Older | 2
  Subjects perception of age at Month 3: 1-5 Years Younger | 12
  Subjects perception of age at Month 3: 6-10 Years Younger | 8
  Subjects perception of age at Month 3: 11-15 Years Younger | 3
  Subjects perception of age at Month 3: 16+ Years Younger | 1
  Subjects perception of age at Month 3: Returned to Baseline | 0
  Subjects perception of age at Month 6: number analyzed (Participants) | 26
  Subjects perception of age at Month 6: Same or Older | 2
  Subjects perception of age at Month 6: 1-5 Years Younger | 12
  Subjects perception of age at Month 6: 6-10 Years Younger | 10
  Subjects perception of age at Month 6: 11-15 Years Younger | 0
  Subjects perception of age at Month 6: 16+ Years Younger | 0
  Subjects perception of age at Month 6: Returned to Baseline | 2
  Subjects perception of age at Month 9: number analyzed (Participants) | 25
  Subjects perception of age at Month 9: Same or Older | 2
  Subjects perception of age at Month 9: 1-5 Years Younger | 11
  Subjects perception of age at Month 9: 6-10 Years Younger | 7
  Subjects perception of age at Month 9: 11-15 Years Younger | 2
  Subjects perception of age at Month 9: 16+ Years Younger | 0
  Subjects perception of age at Month 9: Returned to Baseline | 3
  Subjects perception of age Month 12: number analyzed (Participants) | 25
  Subjects perception of age Month 12: Same or Older | 2
  Subjects perception of age Month 12: 1-5 Years Younger | 12
  Subjects perception of age Month 12: 6-10 Years Younger | 8
  Subjects perception of age Month 12: 11-15 Years Younger | 0
  Subjects perception of age Month 12: 16+ Years Younger | 0
  Subjects perception of age Month 12: Returned to Baseline | 3

5. Other Pre Specified Outcome: Number of Participants With Specific Site Treatment Responses
Description: Site treatment response reported by subject on diary day 0-14 post initial injection and touch-up injections
Time Frame: Day 14
Population: Total number of subjects that reported symptom
Measure: Count of Participants; unit: Participants
Arm/Group | JUVÉDERM VOLUMA™ XC
Number analyzed (Participants) | 30
Participants
  Tenderness/Pain: number analyzed (Participants) | 21
  Tenderness/Pain: Mild | 17
  Tenderness/Pain: Moderate | 3
  Tenderness/Pain: Severe | 1
  Swelling: number analyzed (Participants) | 17
  Swelling: Mild | 17
  Swelling: Moderate | 0
  Swelling: Severe | 0
  Lumps/Bumps: number analyzed (Participants) | 9
  Lumps/Bumps: Mild | 7
  Lumps/Bumps: Moderate | 1
  Lumps/Bumps: Severe | 1
  Bruising: number analyzed (Participants) | 8
  Bruising: Mild | 8
  Bruising: Moderate | 0
  Bruising: Severe | 0
  Redness: number analyzed (Participants) | 8
  Redness: Mild | 7
  Redness: Moderate | 1
  Redness: Severe | 0
  Itching: number analyzed (Participants) | 4
  Itching: Mild | 3
  Itching: Moderate | 1
  Itching: Severe | 0
  Headache: number analyzed (Participants) | 10
  Headache: Mild | 7
  Headache: Moderate | 3
  Headache: Severe | 0
  Jaw Pain/Tension: number analyzed (Participants) | 11
  Jaw Pain/Tension: Mild | 7
  Jaw Pain/Tension: Moderate | 4
  Jaw Pain/Tension: Severe | 0

ADVERSE EVENTS:
Time Frame: Baseline, Month 1, Month 3, Month 6, Month 9, and Month 12
Arm/Group | JUVÉDERM VOLUMA™ XC
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 1/30
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JUVÉDERM VOLUMA™ XC (N=30)
Unexpected Swelling (Skin and subcutaneous tissue disorders) | 1 (1) — Subject experienced unexpected swelling 28 days post injection. Device was removed immediately.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-08-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT02437903/Prot_SAP_000.pdf
  • Informed Consent Form (2015-08-13): https://cdn.clinicaltrials.gov/large-docs/03/NCT02437903/ICF_001.pdf